CLINICAL TRIAL: NCT06998953
Title: Social Isolation But Not Deprivation Involved in Employment Status After Bariatric Surgery.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0005_CHIRURGIE BAR
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Bariatric Surgery; Weight Loss; Employment; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looked at how bariatric surgery (weight-loss surgery) affects people's chances of getting a job, especially in a low-income area. Researchers followed 133 patients (mostly women, average age 45) about 2 years after their surgery. Most had a type of surgery called sleeve gastrectomy and lost a significant amount of weight.

They found that 19 people got a job after surgery, but 3 also became unemployed. People who were already employed before surgery had better results on satisfaction and well-being scores. Interestingly, finding a new job after surgery wasn't linked to weight loss, age, or sex. Also, being poor (measured by the EPICES score) didn't affect employment outcomes. However, people who felt more socially isolated were less likely to lose weight successfully.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent bariatric surgery (mainly sleeve gastrectomy).
* Follow-up duration of approximately 2.3 ± 0.1 years after surgery.
* Residing in a deprived area (context of the study).
* Adults (participants were aged between 18 and 67 years).

Exclusion Criteria:

* Patients who did not undergo bariatric surgery.
* Missing or incomplete data (e.g., unanswered questionnaires).
* Patients outside the follow-up period (less or more than 2.3 years post-surgery).
* Possibly: Minors (<18 years old).

Ages: 18 Years to 67 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults who underwent bariatric surgery, predominantly sleeve gastrectomy, in a socioeconomically deprived area. Participants were selected retrospectively and evaluated at an average of 2.3 years post-surgery. The group included 133 individuals, with a majority being women (approximately 88%), and an average age of 45 years (range: 19-67 years). All participants completed standardized questionnaires assessing deprivation (EPICES score), quality of life and social factors (BAROS score), and satisfaction with outcomes. The population is characterized by severe obesity prior to surgery (mean BMI of 42.7 kg/m²).
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in employment status after bariatric surgery | January 2020 - June 2020

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France